CLINICAL TRIAL: NCT06871982
Title: Norms Re-education to Promote Engagement in Parent-based Interventions: A Type 1 Implementation-effectiveness Trial
Brief Title: Norms Re-education to Promote Engagement in Parent-based Interventions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola Marymount University (Other)
Collaborators: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01AA030904-01 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Underage Drinking
MeSH Terms: conditions — Underage Drinking | interventions — 5-brom-3-(ortho-chlorphenyl)-1-(4-(4-phenyl-1-piperazinyl)butyl)indazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PNF+ PBI (Experimental): This intervention involves an interactive app that delivers six personalized normative feedback quizzes. Based on quiz responses, the app provides tailored videos and readings that address parents' misperceptions about student drinking and offer strategies to reduce alcohol-related risks. The app also includes a resource library and generates customized reading lists through the quizzes.
  Interventions: Behavioral: PNF+ PBI
- SNMC+ PBI (Experimental): This intervention consists of a series of six structured communications that present risk-reducing normative facts about alcohol use. Each communication includes a specific tip designed to guide parents in effectively discussing alcohol-related risks and establishing constructive conversations with their student.
  Interventions: Behavioral: SNMC+ PBI
- PH+ PBI (Active Comparator): This intervention provides a digital version of the Parent Handbook, which contains comprehensive psychoeducational content on alcohol-related risks, effective communication strategies, and practical guidelines for reducing underage drinking. The Handbook is designed to be reviewed at the parent's own pace, offering a thorough resource for managing alcohol-related issues.
  Interventions: Behavioral: PH+ PBI
- No Intervention (No Intervention): In the control condition, no parent-based intervention content is provided.

INTERVENTIONS:
Behavioral: PNF+ PBI — Parents of participating students assigned to the PNF+ PBI condition will receive an email invitation to sign up for a Parent-Based Intervention app. This app features six personalized normative feedback (PNF) quizzes and provides tailored videos and readings based on responses to these quizzes. Parents will create an account and complete the first PNF quiz, after which they will immediately receive their initial set of tailored content. They can then explore additional app content at their convenience, including access to five more quizzes that will yield further customized reading lists and access to a general resource library. For approximately six weeks, parents will receive weekly app notifications and email reminders alerting them to additional unengaged content (e.g., PNF quizzes, readings). Parents in this condition will maintain access to the app throughout their student's first year of college.
  Arms: PNF+ PBI
Behavioral: SNMC+ PBI — Parents of participating students randomized to this condition will receive a series of 6 emails (delivered weekly) in August and September. Each email will include risk-reducing normative facts and a relevant tip for communicating with students about alcohol-related risks.
  Arms: SNMC+ PBI
Behavioral: PH+ PBI — Parents of participating students randomized to this condition will receive an email introducing the PBI including a link to access the Handbook online. Parents can explore the Handbook at their own pace.
  Other Names: Digitized Parent Handbook
  Arms: PH+ PBI

SUMMARY:
A randomized controlled trial (RCT) will be conducted to evaluate both the short-term and long-term efficacy of innovative, incentive-free parent-based interventions (PBIs) designed to reduce underage drinking on college campuses. Although the current NIAAA-recommended Parent Handbook has shown modest effects, our preliminary work suggests that combining personalized normative feedback (PNF) delivered through a social media-inspired app with psychoeducational content can effectively decrease alcohol-related risk. In this large, multi-site trial with 2,040 first-year students, we will examine the short- and long-term effects of the experimental app-based PNF program (PNF+ PBI) compared to an email-based social norms marketing campaign (SNMC+ PBI), the Parent Handbook (PH+ PBI), and an assessment-only control on alcohol use and consequences (primary outcomes). Parent alcohol approval and communication will also be assessed as potential mediators of intervention effects (secondary outcomes). The researchers hypothesize that students whose parents receive PNF+ and SNMC+ PBIs will report lower levels of alcohol use and fewer alcohol-related consequences compared to those whose parents receive PH+ PBI or no intervention. It is also expected that parental approval will be lower and alcohol-related communication will be higher in these two experimental conditions, relative to PH+ PBI and no intervention.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) will be conducted to evaluate the feasibility and efficacy of innovative, incentive-free parent-based interventions (PBIs) designed to reduce underage drinking on college campuses. Incoming first-year students will be invited to complete an online baseline survey during the summer prior to matriculation to assess alcohol use and related behaviors. An automated randomizer embedded in the survey will assign students (and thus their parents) to one of four conditions: an experimental app-based personalized normative feedback program (PNF+ PBI), an email-based social norms marketing campaign (SNMC+ PBI), the NIAAA-recommended Parent Handbook (PH+ PBI), or an assessment-only control group. Parents in the PBI conditions will receive access to their assigned program in July or August (immediately following their students completion of the baseline survey). Students will complete a total of four surveys: the baseline assessment and three follow-up surveys at one month, six months, and twelve months post-matriculation. The researchers hypothesize that students whose parents are assigned to the experimental app-based PNF and email-based SNMC conditions will report lower alcohol use and fewer alcohol-related consequences compared to those whose parents receive the Parent Handbook or no intervention. In addition, it is expected that these experimental conditions will yield lower parental alcohol approval and higher levels of alcohol-related communication, which will serve as potential mediators of the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* LMU/Lehigh incoming first-year college student who is17-20 years of age
* Parent/legal guardian with an email address on file with the university
* A United States resident
* Provide informed consent/assent

Exclusion Criteria:

* Younger than 17 or older than 20 years of age
* Not an incoming first-year college students at LMU/Lehigh
* Parent or legal guardian does not have an email address on file with the university
* Not residents of the United States
* Did not provide informed consent/assent

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2040 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline Daily Drinking from Baseline to 1 Month Post Intervention | baseline, 3 months
  Self-reported number of drinks consumed during an average week in the past 30 days.
Change in Baseline Daily Drinking from Baseline to 7 Months Post Intervention | baseline, 7 months
  Self-reported number of drinks consumed during an average week in the past 30 days.
Change in Baseline Daily Drinking from Baseline to 12 Months Post Intervention | baseline, 12 months
  Self-reported number of drinks consumed during an average week in the past 30 days.
Change in Peak Drinking from Baseline to 1 Month Post Intervention | baseline, 1 month
  Self-reported max number of drinks consumed on a single occasion in the past 30 days.
Change in Peak Drinking from Baseline to 7 Months Post Intervention | baseline, 7 months
  Self-reported max number of drinks consumed on a single occasion in the past 30 days.
Change in Peak Drinking from Baseline to 12 Months Post Intervention | baseline, 12 months
  Self-reported max number of drinks consumed on a single occasion in the past 30 days.
Change in Heavy Episodic Drinking from Baseline to 1 Month Post Intervention | baseline, 1 month
  Self-reported number of times 4/5 drinks (female/male) were consumed in a 2-hour period in the past 30 days
Change in Heavy Episodic Drinking from Baseline to 7 Months Post Intervention | baseline, 7 months
  Self-reported number of times 4/5 drinks (female/male) were consumed in a 2-hour period in the past 30 days
Change in Heavy Episodic Drinking from Baseline to 12 Months Post Intervention | baseline, 12 months
  Self-reported number of times 4/5 drinks (female/male) were consumed in a 2-hour period in the past 30 days
Change in High Intensity Drinking from Baseline to 1 Month Post Intervention | baseline, 1 month
  Self-reported number of times 8/10 drinks (female/male) were consumed on a single occasion in the past 30 days
Change in High Intensity Drinking from Baseline to 7 Months Post Intervention | baseline, 7 months
  Self-reported number of times 8/10 drinks (female/male) were consumed on a single occasion in the past 30 days
Change in High Intensity Drinking from Baseline to 12 Months Post Intervention | baseline, 12 months
  Self-reported number of times 8/10 drinks (female/male) were consumed on a single occasion in the past 30 days
Change in Alcohol-Related Consequences from Baseline to 1 Month Post Intervention | baseline, 1 month
  Self-reported number of alcohol-related consequences in the past 30 days.
Change in Alcohol-Related Consequences from Baseline to 7 Months Post Intervention | baseline, 7 months
  Self-reported number of alcohol-related consequences in the past 30 days.
Change in Alcohol-Related Consequences from Baseline to 12 Months Post Intervention | baseline, 12 months
  Self-reported number of alcohol-related consequences in the past 30 days.

SECONDARY OUTCOMES:
Change in Perceived Parental Approval of Underage Drinking from Baseline to 1 Month Post Intervention | baseline, 1 month
  Self-reported number of drinks parent would permit student to drink in the next year.
Change in Perceived Parental Approval of Underage Drinking from Baseline to 7 Months Post Intervention | baseline, 7 months
  Self-reported number of drinks parent would permit student to drink in the next year.
Change in Perceived Parental Approval of Underage Drinking from Baseline to 12 Months Post Intervention | baseline, 12 months
  Self-reported number of drinks parent would permit student to drink.
Change in Perceived Frequency of Parent Communication from Baseline to 1 Month Post Intervention | baseline, 1 month
  Self-reported frequency of parent communication in the past 3 months.
Change in Perceived Frequency of Parent Communication from Baseline to 7 Months Post Intervention | baseline, 7 months
  Self-reported frequency of parent communication in the past 3 months.
Change in Perceived Frequency of Parent Communication from Baseline to 12 Months Post Intervention | baseline, 12 months
  Self-reported frequency of parent communication in the past 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola Marymount, Los Angeles, California, United States